CLINICAL TRIAL: NCT00430716
Title: A MULTINATIONAL, MULTICENTRE, RANDOMIZED, PARALLEL GROUP, DOUBLE-BLIND STUDY TO ASSESS THE EFFICACY AND SAFETY OF 1MG, 5MG AND 20 MG TID OF ORAL SILDENAFIL IN THE TREATMENT OF SUBJECTS AGED 18 YEARS AND OVER WITH PULMONARY ARTERIAL HYPERTENSION (PAH)
Brief Title: To Assess The Efficacy and Safety Of Oral Sildenafil in the Treatment of Pulmonary Arterial Hypertension.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was terminated at the recommendation of an independent Data Monitoring Committee. The decision was not based on any safety concerns.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A1481244; 2006-006748-76 (EudraCT Number)
Record Dates: First submitted 2007-01-31; First posted 2007-02-02 (Estimated); Results first posted 2011-05-17 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sildenafil High dose (Experimental)
  Interventions: Drug: Sildenafil citrate
- Sildenafil Low dose (Experimental)
  Interventions: Drug: Sildenafil citrate
- Sildenafil medium dose (Experimental)
  Interventions: Drug: Sildenafil citrate
- Sildenafil - Open label Phase (Experimental): Open label extension from week 12 to week 24.
  Interventions: Drug: Sildenafil citrate

INTERVENTIONS:
Drug: Sildenafil citrate — oral, 20 mg, tid
  Arms: Sildenafil High dose
Drug: Sildenafil citrate — oral 1 mg, tid
  Arms: Sildenafil Low dose
Drug: Sildenafil citrate — oral 5 mg, tid
  Arms: Sildenafil medium dose
Drug: Sildenafil citrate — oral 20 mg, tid
  Arms: Sildenafil - Open label Phase

SUMMARY:
To demonstrate a dose response for 1 mg, 5 mg and 20 mg TID oral sildenafil for the treatment of subjects with PAH.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with PAH (i.e. IPAH or secondary to connective tissue disease or with surgical repair of ASD, VSD, PDA, aorto-pulmonary window) whose baseline six minute walk test distance is >/= 100 m and </= 450 m.
* Subjects with a mean pulmonary artery pressure of >/= 25 mmHg and a pulmonary artery wedge pressure of </= 15 mmHg at rest via right heart catheterization performed within 12 weeks prior to randomization.

Exclusion Criteria:

* Subjects whose 6 Minute Walk Distance may be limited by conditions other than PAH related dyspnoea or fatigue, e.g. claudication from vascular insufficiency or significant arthritis.
* Subjects who are currently receiving any forms of chronic treatment for PAH such as prostacyclin, PDE-5 inhibitors, endothelin-receptor antagonists, nitrates or nitric oxide donors (e.g. arginine supplement, nicorandil) in any form, protease inhibitors such as ritonavir and saquinavir, ketoconazole, itraconazole, and alpha blockers. Subjects previously receiving any of these drugs must have stopped use for a period of at least 1 month prior to screening, except in the case of bosentan or prostacyclin (3 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-04-08 (Actual); Primary Completion 2010-05-25 (Actual); Study Completion 2010-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (15):
  - Arizona Pulmonary Specialists, LTD, Phoenix, Arizona
  - Medical College of Georgia, Augusta, Georgia
  - Atlanta Institute for Medical Research, Inc., Decatur, Georgia
  - Chicago Heart Institute, Elk Grove Village, Illinois
  - The Care Group, LLC, Indianapolis, Indiana
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Mid Carolina Cardiology, Charlotte, North Carolina
  - Presbyterian Hospital, Charlotte, North Carolina
  - Baylor College of Medicine Pulmonary Section, Houston, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - University of Utah Sciences Center, Salt Lake City, Utah
  - CJW Chippenham Medical Center, Richmond, Virginia
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
  - Virginia Cardiovascular Specialists, Richmond, Virginia
  - Cardiovascular Associates of Virginia, Richmond, Virginia
- Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven, Belgium
- Brazil (2):
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo
- Bulgaria (2):
  - Peta mnogoprofilna bolnitsa za aktivno lechenie, Klinika po kardiologia, Sofia
  - Mnogoprofilna bolnitsa za aktivno lechenie i speshna meditsina "N.I.Pirogov", Sofia
- China (2):
  - Beijing Shijitan Hospital, Beijing
  - Shanghai Pulmonology Hospital, Shanghai
- Attikon Hospital, Haidari, Athens, Greece
- India (5):
  - Care Hospital, The Institute of Medical Sciences, Hyderabad, Andhra Pradesh
  - Mehta Hospital & Cardiopulmonary Care Center, Ahmedabad, Gujarat
  - Bankers Heart Institute, Vadodara, Gujarat
  - St. John's Medical College Hospital, Bangalore, Karnataka
  - Metro Multispeciality Hospital, Noida, Uttar Pradesh
- Italy (2):
  - IRCCS Policlinico San Matteo, Pavia
  - Unita' di Ipertensione Polmonare, Dipartimento di Scienze Respiratorie e Cardiovascolari, Roma
- P. Stradins Clinical University Hospital / Latvian Centre of Cardilogy, Riga, Latvia
- National Heart Institute, Kuala Lumpur, Malaysia
- Netherlands (2):
  - VU Medisch Centrum / afdeling Longziekten, Amsterdam
  - Erasmus MC, Rotterdam
- Philippines (2):
  - Philippine General Hospital, Manila
  - Philippine Heart Center, Quezon City
- Poland (2):
  - Krakowski Szpital Specjalistyczny Im. Jana Pawla II w Krakowie, Krakow
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Slaskie Centrum Chorob Serca, Zabrze
- Romania (2):
  - Spitalul Clinic de Boli Infectioase si Pneumoftiziologie Dr. Victor Babes, Timișoara, Timiș County
  - Spitalul Clinic de Pneumoftiziologie, Iași
- Scientific Center of Cardiovascular surgery n.a. A.N.Bakoulev RAMS, Moscow, Russia
- Thailand (2):
  - Division of Rheumatology Allergy and Immunology, Department of Medicine, Faculty of Medicine, Amphoe Mueang, Changwat Khon Kaen
  - Department of Medicine,, Bangkok
- United Kingdom (2):
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Room 224A Sir William Leech Centre, Newcastle upon Tyne, TYNE and WEAR

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Vizza CD, Sastry BK, Safdar Z, Harnisch L, Gao X, Zhang M, Lamba M, Jing ZC. Efficacy of 1, 5, and 20 mg oral sildenafil in the treatment of adults with pulmonary arterial hypertension: a randomized, double-blind study with open-label extension. BMC Pulm Med. 2017 Feb 23;17(1):44. doi: 10.1186/s12890-017-0374-x. PMID 28228114
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481244&StudyName=To%20Assess%20The%20Efficacy%20and%20Safety%20Of%20%20Oral%20Sildenafil%20in%20the%20Treatment%20of%20Pulmonary%20Arterial%20Hypertension.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sildenafil 1 mg: Sildenafil 1 milligram (mg) tablet taken orally 3 times a day (TID) for first 12 weeks (double blind treatment phase of the study) and placebo matched to 20 mg. For a further 12 weeks (open label extension phase), participants received sildenafil 20 mg tablets TID.
- Sildenafil 5 mg: Sildenafil 5 mg tablet taken orally TID for first 12 weeks (double blind treatment phase of the study) and placebo matched to 20 mg. For a further 12 weeks (open label extension phase), participants received sildenafil 20 mg tablets TID.
- Sildenafil 20 mg: Sildenafil 20 mg tablet taken orally TID throughout the study and placebo matched to 1 and 5 mg during first 12 weeks (double blind treatment phase).
Period: Double Blind Phase
Arm/Group | Sildenafil 1 mg | Sildenafil 5 mg | Sildenafil 20 mg
Started | 42 | 43 | 45
Treated | 41 | 43 | 45
Completed | 36 | 38 | 39
Not Completed | 6 | 5 | 6
Not completed — Death | 1 | 0 | 0
Not completed — No longer willing to participate | 2 | 1 | 1
Not completed — Other | 0 | 2 | 0
Not completed — Study terminated by sponsor | 1 | 1 | 2
Not completed — Adverse Event | 1 | 1 | 3
Not completed — Not treated | 1 | 0 | 0
Period: Open Label Phase
Arm/Group | Sildenafil 1 mg | Sildenafil 5 mg | Sildenafil 20 mg
Started | 36 | 38 | 39
Completed | 27 | 31 | 32
Not Completed | 9 | 7 | 7
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — No longer willing to participate | 0 | 1 | 1
Not completed — Other | 3 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Study terminated by sponsor | 4 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil 1 mg | Sildenafil 5 mg | Sildenafil 20 mg | Total
Number analyzed (Participants) | 41 | 43 | 45 | 129
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.5 (16.5) | 44.4 (17.4) | 46.4 (17.7) | 44.5 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 33 | 26 | 87
  Male | 13 | 10 | 19 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Total Distance Walked During 6-Minute Walk Test (6MWT) at Week 12
Description: 6 MWT was the distance that a participant could walk in 6 minutes. Participants were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed. Continuous pulse oximetry was conducted during the test for safety.
Time Frame: Baseline and Week 12
Population: Intention to Treat (ITT population) included all participants who were randomized to study treatment and received at least 1 dose of study medication. If participant had missing value at any visit, last observation carried forward (LOCF) method of imputation was used.
Measure: Mean (95% Confidence Interval); unit: Meters
Arm/Group | Sildenafil 1 mg | Sildenafil 5 mg | Sildenafil 20 mg
Number analyzed (Participants) | 41 | 40 | 42
Meters | 14.21 [0.41 to 28.00] | 40.75 [25.16 to 56.34] | 38.36 [23.77 to 52.94]
Statistical Analysis 1: Comparison: Sildenafil 1 mg vs Sildenafil 20 mg; An analysis of variance (ANOVA) model followed by the Williams trend test (one-sided, at the 2.5% level of significance) was used. The Williams trend test firstly determined if there was a significant downward trend in response for the descending doses, and then subsequently determined the highest dose that was statistically inferior to 20 mg (known to be an effective dose of sildenafil). A corresponding 97.5% lower confidence limit for the difference was presented; Test type: Superiority or Other; p = 0.011, ANOVA; Mean Difference (Net) = 24.15, 97.5% CI 1-sided [lower limit 3.37]
Statistical Analysis 2: Comparison: Sildenafil 5 mg vs Sildenafil 20 mg; ANOVA model followed by the Williams trend test (one-sided, at the 2.5% level of significance) was used. The Williams trend test firstly determined if there was a significant downward trend in response for the descending doses, and then subsequently determined the highest dose that was statistically inferior to 20 mg (known to be an effective dose of sildenafil). A corresponding 97.5% lower confidence limit for the difference was presented; Test type: Superiority or Other; p = 0.545, ANOVA; Mean Difference (Net) = -1.17, 97.5% CI 1-sided [lower limit -21.48]

2. Secondary Outcome: Change From Baseline in Mean Pulmonary Arterial Pressure (mPAP) at Week 12
Description: mPAP was measured using a pressure transducer positioned at the mid-axillary line.
Time Frame: Baseline and Week 12
Population: ITT population included all participants who were randomized to study treatment and received at least 1 dose of study medication. If participant had missing value at any visit, LOCF method of imputation was used.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Sildenafil 1 mg | Sildenafil 5 mg | Sildenafil 20 mg
Number analyzed (Participants) | 33 | 33 | 34
mmHg | -1.73 [-5.99 to 2.54] | -3.44 [-5.87 to -1.00] | -3.29 [-6.05 to -0.52]
Statistical Analysis 1: Comparison: Sildenafil 1 mg vs Sildenafil 20 mg; The analysis of change from baseline in week 12 mean PAP used Analysis of Covariance (ANCOVA), with etiology and baseline walking distance category (<325m or >=325m) and baseline score as the covariates. The mean difference and corresponding two-sided 95% CI for the comparisons of sildenafil 20 mg against the lower sildenafil dose (1 mg) was presented along with the p-value for the test; Test type: Superiority or Other; p = 0.278, ANCOVA; Mean Difference (Net) = -2.51, 95% CI 2-sided [-7.07 to 2.05]
Statistical Analysis 2: Comparison: Sildenafil 5 mg vs Sildenafil 20 mg; The analysis of change from baseline in week 12 mean PAP used ANCOVA, with etiology and baseline walking distance category (<325m or >=325m) and baseline score as the covariates. The mean difference and corresponding two-sided 95% CI for the comparisons of sildenafil 20 mg against the lower sildenafil dose (5 mg) was presented along with the p-value for the test; Test type: Superiority or Other; p = 0.846, ANCOVA; Mean Difference (Net) = -0.44, 95% CI 2-sided [-4.98 to 4.09]

3. Secondary Outcome: Number of Participants With Clinical Worsening
Description: Clinical worsening was defined as death; or lung transplantation; or hospitalization due to pulmonary hypertension; or initiation of prostacyclin therapy; or initiation of endothelin receptor antagonist therapy. (PAH=pulmonary arterial hypertension) Due to very low number of events of clinical worsening reported, the median days to clinical worsening could not be estimated.
Time Frame: Baseline through Week 12
Population: ITT population for clinical worsening included all participants who had been randomized to study treatment and received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Sildenafil 1 mg | Sildenafil 5 mg | Sildenafil 20 mg
Number analyzed (Participants) | 41 | 43 | 45
Participants
  death | 1 | 1 | 0
  lung transplantation | 0 | 0 | 0
  hospitalisation due to pulmonary hypertension | 1 | 0 | 2
  PAH deterioration requiring therapy | 0 | 0 | 0
  receptor antagonist therapy | 0 | 1 | 0

4. Secondary Outcome: Number of Participants With Change From Baseline in PAH Criteria for Functional Capacity and Therapeutic Class at Week 12
Description: Pulmonary arterial hypertension (PAH) Criteria for WHO Class: Class I (Participants without resulting limitation of physical activity);Class II (Participants with slight limitation of physical activity though comfortable at rest);Class III (Participants with marked limitation of physical activity,though comfortable at rest);Class IV(Participants with inability to carry out any physical activity without symptoms,manifest signs of right heart failure; dyspnoea and/or fatigue may even be present at rest; and discomfort is increased by any physical activity).
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Sildenafil 1 mg | Sildenafil 5 mg | Sildenafil 20 mg
Number analyzed (Participants) | 41 | 43 | 45
Participants
  Worsened 2 Classes | 0 | 0 | 0
  Worsened 1 Class | 1 | 3 | 2
  No Change | 35 | 27 | 35
  Improved 1 Class | 4 | 10 | 6
  Improved 2 Classes | 1 | 0 | 0
  Missing | 0 | 3 | 2
Statistical Analysis 1: Comparison: Sildenafil 1 mg vs Sildenafil 20 mg; The analysis of the week 12 PAH functional class was done with etiology, baseline walking distance category (<325m or >=325m) and baseline score as the covariates.The odds ratio and corresponding two-sided 95% CI for the odds ratio for the treatment comparisons was presented along with the p-value for the tests; Test type: Superiority or Other; p = 0.448, Regression, Logistic; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.50 to 4.78]
Statistical Analysis 2: Comparison: Sildenafil 5 mg vs Sildenafil 20 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.897, Regression, Logistic; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.35 to 3.32]

5. Secondary Outcome: Change From Baseline in B-Type Natriuretic Peptide (BNP) at Week 12
Description: BNP is a non-invasive biomarker and an indicator of progression of PAH/ right ventricular dysfunction in participants with PAH.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Sildenafil 1 mg | Sildenafil 5 mg | Sildenafil 20 mg
Number analyzed (Participants) | 38 | 39 | 42
pg/mL | -6.28 [-80.75 to 68.19] | -53.46 [-99.98 to -6.94] | -97.42 [-161.45 to -33.39]
Statistical Analysis 1: Comparison: Sildenafil 1 mg vs Sildenafil 20 mg; ANCOVA method was used with etiology, baseline walking distance category (<325m or >=325m) and baseline score as the covariates. The mean difference and corresponding two-sided 95% CI for the comparisons of sildenafil 20 mg against the lower sildenafil dose (1 mg) was presented along with the p-value for the test; Test type: Superiority or Other; p = 0.005, ANCOVA; Mean Difference (Net) = -104.80, 95% CI 2-sided [-177.44 to -32.16]
Statistical Analysis 2: Comparison: Sildenafil 5 mg vs Sildenafil 20 mg; ANCOVA method was used with etiology, baseline walking distance category (<325m or >=325m) and baseline score as the covariates. The mean difference and corresponding two-sided 95% CI for the comparisons of sildenafil 20 mg against the lower sildenafil dose (5 mg) was presented along with the p-value for the test; Test type: Superiority or Other; p = 0.496, ANCOVA; Mean Difference (Net) = -25.00, 95% CI 2-sided [-97.50 to 47.50]

6. Secondary Outcome: Change From Baseline in Pro-BNP at Week 12
Description: Pro- BNP which is a precursor of BNP, is a non-invasive biomarker and an indicator of progression of PAH / RV dysfunction in participants with PAH.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Sildenafil 1 mg | Sildenafil 5 mg | Sildenafil 20 mg
Number analyzed (Participants) | 39 | 40 | 43
pg/mL | -111.53 [-507.68 to 284.63] | -306.76 [-523.82 to -89.70] | -428.54 [-676.74 to -180.34]
Statistical Analysis 1: Comparison: Sildenafil 1 mg vs Sildenafil 20 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.009, ANCOVA; Mean Difference (Net) = -462.12, 95% CI 2-sided [-807.53 to -116.71]
Statistical Analysis 2: Comparison: Sildenafil 5 mg vs Sildenafil 20 mg; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.414, ANCOVA; Median Difference (Net) = -141.45, 95% CI 2-sided [-483.48 to 200.58]

7. Secondary Outcome: Change From Baseline in TAPSE Measurement at Week 12
Description: Tricuspid annular plane systolic excursion (TAPSE) was measured as the total displacement of the tricuspid annulus in cm from end diastole to end systole.TAPSE is an indicator of progression of PAH /right ventricular dysfunction.
  The baseline data for 33 participants were measured incorrectly and the results from the 33 participants (both baseline and post-baseline) were excluded from the analysis.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Sildenafil 1 mg | Sildenafil 5 mg | Sildenafil 20 mg
Number analyzed (Participants) | 32 | 29 | 28
cm | 0.08 [-0.04 to 0.19] | 0.17 [0.05 to 0.29] | -0.02 [-0.15 to 0.10]
Statistical Analysis 1: Comparison: Sildenafil 1 mg vs Sildenafil 20 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.890, ANCOVA; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.17 to 0.15]
Statistical Analysis 2: Comparison: Sildenafil 5 mg vs Sildenafil 20 mg; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.124, ANCOVA; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.29 to 0.04]

8. Secondary Outcome: Change From Baseline in BORG Dyspnoea Score at Week 12
Description: BORG dyspnoea scale is a 10-point scale where following scores stands for severity of dyspnoea: 0 (no breathlessness at all); 0.5 (very very slight [just noticeable]); 1 (very slight); 2 (slight breathlessness); 3 (moderate); 4 (some what severe); 5 (severe breathlessness); 7 (very severe breathlessness); 9 (very very severe [almost maximum] and 10 (maximum).
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Sildenafil 1 mg | Sildenafil 5 mg | Sildenafil 20 mg
Number analyzed (Participants) | 41 | 40 | 42
Units on a scale | -0.28 [-0.76 to 0.20] | -0.89 [-1.35 to -0.43] | -0.43 [-0.94 to 0.08]
Statistical Analysis 1: Comparison: Sildenafil 1 mg vs Sildenafil 20 mg; A stratified Wilcoxon test (Van-Elteren) was used. The stratified median difference and corresponding two-sided 95% CI (calculated using the Hodges-Lehmann estimator) was presented along with the p-value for the test; Test type: Superiority or Other; p = 0.382, Wilcoxon (Van-Elteren); Median Difference (Net) = 0.00, 95% CI 2-sided [-1.00 to 0.00]
Statistical Analysis 2: Comparison: Sildenafil 5 mg vs Sildenafil 20 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.141, Wilcoxon (Van-Elteren); Mean Difference (Net) = 0.00, 95% CI 2-sided [0.00 to 1.00]

ADVERSE EVENTS:
Time Frame: 24 Weeks
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sildenafil 1 mg | Sildenafil 5 mg | Sildenafil 20 mg
All-Cause Mortality (participants affected / at risk) | 1/41 | 1/43 | 0/45
Serious Adverse Events (participants affected / at risk) | 6/41 | 3/43 | 5/45
Other Adverse Events (participants affected / at risk) | 21/41 | 22/43 | 22/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil 1 mg (N=41) | Sildenafil 5 mg (N=43) | Sildenafil 20 mg (N=45)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 — Double Blind Phase
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 — Double Blind Phase
Cor pulmonale (Cardiac disorders) | 1 | 0 | 0 — Double Blind Phase
Right ventricular failure (Cardiac disorders) | 0 | 0 | 1 — Double Blind Phase
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 — Double Blind Phase
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 — Double Blind Phase
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 — Double Blind Phase
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 — Double Blind Phase
Pneumonia (Infections and infestations) | 1 | 0 | 0 — Double Blind Phase
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 — Double Blind Phase
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — Double Blind Phase
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — Double Blind Phase
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 — Open Label Phase
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 — Open Label Phase
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 — Open Label Phase
Cor pulmonale (Cardiac disorders) | 1 | 0 | 0 — Open Label Phase
Right ventricular failure (Cardiac disorders) | 0 | 0 | 2 — Open Label Phase
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 — Open Label Phase
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 — Open Label Phase
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 — Open Label Phase
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 — Open Label Phase
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 — Open Label Phase
Pneumonia (Infections and infestations) | 1 | 0 | 0 — Open Label Phase
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 — Open Label Phase
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 — Open Label Phase
Blood electrolytes abnormal (Investigations) | 1 | 0 | 0 — Open Label Phase
International normalised ratio increased (Investigations) | 1 | 0 | 0 — Open Label Phase
Weight increased (Investigations) | 0 | 0 | 1 — Open Label Phase
Syncope (Nervous system disorders) | 0 | 1 | 0 — Open Label Phase
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Open Label Phase
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 — Open Label Phase
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — Open Label Phase
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 — Open Label Phase
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — Open Label Phase
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil 1 mg (N=41) | Sildenafil 5 mg (N=43) | Sildenafil 20 mg (N=45)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2 — Double Blind Phase
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 — Double Blind Phase
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 — Double Blind Phase
Cyanosis (Cardiac disorders) | 0 | 1 | 0 — Double Blind Phase
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0 — Double Blind Phase
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0 — Double Blind Phase
Tachycardia (Cardiac disorders) | 1 | 0 | 0 — Double Blind Phase
Hereditary haemorrhagic telangiectasia (Congenital, familial and genetic disorders) | 0 | 0 | 1 — Double Blind Phase
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 — Double Blind Phase
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 — Double Blind Phase
Conjunctivitis (Eye disorders) | 0 | 1 | 0 — Double Blind Phase
Periorbital oedema (Eye disorders) | 1 | 0 | 0 — Double Blind Phase
Photophobia (Eye disorders) | 0 | 1 | 0 — Double Blind Phase
Vision blurred (Eye disorders) | 0 | 1 | 0 — Double Blind Phase
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 — Double Blind Phase
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 — Double Blind Phase
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 — Double Blind Phase
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 — Double Blind Phase
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 — Double Blind Phase
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 — Double Blind Phase
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 — Double Blind Phase
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 — Double Blind Phase
Asthenia (General disorders) | 1 | 1 | 1 — Double Blind Phase
Exercise tolerance decreased (General disorders) | 0 | 0 | 1 — Double Blind Phase
Fatigue (General disorders) | 2 | 1 | 0 — Double Blind Phase
Feeling hot (General disorders) | 0 | 0 | 1 — Double Blind Phase
Medical device pain (General disorders) | 1 | 0 | 0 — Double Blind Phase
Oedema peripheral (General disorders) | 1 | 1 | 2 — Double Blind Phase
Pyrexia (General disorders) | 1 | 1 | 0 — Double Blind Phase
Bronchitis (Infections and infestations) | 1 | 0 | 0 — Double Blind Phase
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 1 — Double Blind Phase
Herpes zoster (Infections and infestations) | 1 | 0 | 0 — Double Blind Phase
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1 — Double Blind Phase
Otitis externa (Infections and infestations) | 1 | 0 | 0 — Double Blind Phase
Rhinitis (Infections and infestations) | 0 | 1 | 0 — Double Blind Phase
Sinusitis (Infections and infestations) | 0 | 1 | 0 — Double Blind Phase
Tinea barbae (Infections and infestations) | 1 | 0 | 0 — Double Blind Phase
Blood potassium decreased (Investigations) | 1 | 0 | 0 — Double Blind Phase
Prostatic specific antigen increased (Investigations) | 0 | 1 | 0 — Double Blind Phase
Weight decreased (Investigations) | 0 | 1 | 0 — Double Blind Phase
Weight increased (Investigations) | 0 | 0 | 1 — Double Blind Phase
White blood cell count decreased (Investigations) | 0 | 1 | 0 — Double Blind Phase
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 — Double Blind Phase
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 — Double Blind Phase
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 — Double Blind Phase
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 — Double Blind Phase
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — Double Blind Phase
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 — Double Blind Phase
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 — Double Blind Phase
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 — Double Blind Phase
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — Double Blind Phase
Dizziness (Nervous system disorders) | 2 | 1 | 1 — Double Blind Phase
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 — Double Blind Phase
Headache (Nervous system disorders) | 1 | 1 | 3 — Double Blind Phase
Lethargy (Nervous system disorders) | 1 | 0 | 0 — Double Blind Phase
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 — Double Blind Phase
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 — Double Blind Phase
Presyncope (Nervous system disorders) | 0 | 1 | 0 — Double Blind Phase
Sciatica (Nervous system disorders) | 1 | 0 | 0 — Double Blind Phase
Anxiety (Psychiatric disorders) | 1 | 0 | 0 — Double Blind Phase
Depression (Psychiatric disorders) | 1 | 0 | 0 — Double Blind Phase
Insomnia (Psychiatric disorders) | 1 | 0 | 0 — Double Blind Phase
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 — Double Blind Phase
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 — Double Blind Phase
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3 — Double Blind Phase
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 — Double Blind Phase
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — Double Blind Phase
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Double Blind Phase
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Double Blind Phase
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — Double Blind Phase
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Double Blind Phase
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 — Double Blind Phase
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Double Blind Phase
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Double Blind Phase
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 — Double Blind Phase
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 — Double Blind Phase
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 — Double Blind Phase
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 — Double Blind Phase
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 — Double Blind Phase
Flushing (Vascular disorders) | 0 | 2 | 1 — Double Blind Phase
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 — Double Blind Phase
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 — Open Label Phase
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 — Open Label Phase
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 — Open Label Phase
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 — Open Label Phase
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 — Open Label Phase
Cyanosis (Cardiac disorders) | 0 | 1 | 0 — Open Label Phase
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0 — Open Label Phase
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 — Open Label Phase
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0 — Open Label Phase
Tachycardia (Cardiac disorders) | 1 | 0 | 0 — Open Label Phase
Hereditary haemorrhagic telangiectasia (Congenital, familial and genetic disorders) | 0 | 0 | 1 — Open Label Phase
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 — Open Label Phase
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 — Open Label Phase
Goitre (Endocrine disorders) | 1 | 0 | 0 — Open Label Phase
Blindness transient (Eye disorders) | 0 | 1 | 1 — Open Label Phase
Conjunctivitis (Eye disorders) | 0 | 1 | 0 — Open Label Phase
Periorbital oedema (Eye disorders) | 1 | 0 | 0 — Open Label Phase
Photophobia (Eye disorders) | 1 | 1 | 0 — Open Label Phase
Vision blurred (Eye disorders) | 1 | 1 | 0 — Open Label Phase
Visual impairment (Eye disorders) | 1 | 0 | 0 — Open Label Phase
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 — Open Label Phase
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 — Open Label Phase
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 — Open Label Phase
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 — Open Label Phase
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 — Open Label Phase
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 — Open Label Phase
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 — Open Label Phase
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 — Open Label Phase
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 — Open Label Phase
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 — Open Label Phase
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 — Open Label Phase
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 — Open Label Phase
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 — Open Label Phase
Asthenia (General disorders) | 1 | 2 | 2 — Open Label Phase
Chest pain (General disorders) | 0 | 2 | 0 — Open Label Phase
Exercise tolerance decreased (General disorders) | 0 | 0 | 1 — Open Label Phase
Fatigue (General disorders) | 3 | 1 | 0 — Open Label Phase
Feeling hot (General disorders) | 0 | 0 | 1 — Open Label Phase
Medical device pain (General disorders) | 1 | 0 | 0 — Open Label Phase
Oedema (General disorders) | 1 | 0 | 0 — Open Label Phase
Oedema peripheral (General disorders) | 1 | 1 | 2 — Open Label Phase
Pyrexia (General disorders) | 2 | 2 | 0 — Open Label Phase
Bronchitis (Infections and infestations) | 1 | 1 | 1 — Open Label Phase
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 1 — Open Label Phase
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 — Open Label Phase
Herpes zoster (Infections and infestations) | 1 | 0 | 0 — Open Label Phase
Infected bites (Infections and infestations) | 0 | 1 | 0 — Open Label Phase
Influenza (Infections and infestations) | 0 | 0 | 1 — Open Label Phase
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1 — Open Label Phase
Nasopharyngitis (Infections and infestations) | 2 | 1 | 3 — Open Label Phase
Otitis externa (Infections and infestations) | 1 | 0 | 0 — Open Label Phase
Rhinitis (Infections and infestations) | 0 | 1 | 0 — Open Label Phase
Sinusitis (Infections and infestations) | 1 | 1 | 0 — Open Label Phase
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 — Open Label Phase
Tinea barbae (Infections and infestations) | 1 | 0 | 0 — Open Label Phase
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 — Open Label Phase
Blood potassium decreased (Investigations) | 2 | 0 | 0 — Open Label Phase
Blood pressure increased (Investigations) | 1 | 0 | 0 — Open Label Phase
Blood urea increased (Investigations) | 0 | 1 | 0 — Open Label Phase
Prostatic specific antigen increased (Investigations) | 0 | 1 | 0 — Open Label Phase
Weight decreased (Investigations) | 1 | 2 | 0 — Open Label Phase
Weight increased (Investigations) | 1 | 0 | 1 — Open Label Phase
White blood cell count decreased (Investigations) | 0 | 1 | 0 — Open Label Phase
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 — Open Label Phase
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 — Open Label Phase
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 — Open Label Phase
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 — Open Label Phase
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 — Open Label Phase
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 — Open Label Phase
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 — Open Label Phase
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 — Open Label Phase
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 — Open Label Phase
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — Open Label Phase
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 — Open Label Phase
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 — Open Label Phase
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 — Open Label Phase
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 — Open Label Phase
Dizziness (Nervous system disorders) | 3 | 2 | 2 — Open Label Phase
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 — Open Label Phase
Head discomfort (Nervous system disorders) | 0 | 0 | 1 — Open Label Phase
Headache (Nervous system disorders) | 2 | 3 | 3 — Open Label Phase
Lethargy (Nervous system disorders) | 1 | 1 | 1 — Open Label Phase
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 — Open Label Phase
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 — Open Label Phase
Presyncope (Nervous system disorders) | 0 | 2 | 0 — Open Label Phase
Sciatica (Nervous system disorders) | 1 | 0 | 0 — Open Label Phase
Syncope (Nervous system disorders) | 0 | 1 | 0 — Open Label Phase
Anxiety (Psychiatric disorders) | 1 | 0 | 0 — Open Label Phase
Depression (Psychiatric disorders) | 1 | 0 | 0 — Open Label Phase
Insomnia (Psychiatric disorders) | 1 | 1 | 0 — Open Label Phase
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 — Open Label Phase
Renal failure (Renal and urinary disorders) | 1 | 0 | 1 — Open Label Phase
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 — Open Label Phase
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 — Open Label Phase
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3 — Open Label Phase
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 — Open Label Phase
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — Open Label Phase
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 — Open Label Phase
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Open Label Phase
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Open Label Phase
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — Open Label Phase
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Open Label Phase
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 — Open Label Phase
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Open Label Phase
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Open Label Phase
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 — Open Label Phase
Butterfly rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 — Open Label Phase
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 — Open Label Phase
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 — Open Label Phase
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 — Open Label Phase
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 — Open Label Phase
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 — Open Label Phase
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 — Open Label Phase
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 — Open Label Phase
Flushing (Vascular disorders) | 0 | 2 | 1 — Open Label Phase
Hypertension (Vascular disorders) | 1 | 0 | 0 — Open Label Phase
Hypotension (Vascular disorders) | 1 | 0 | 1 — Open Label Phase
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 — Open Label Phase

LIMITATIONS AND CAVEATS:
The trial was not designed to demonstrate the equivalence of doses and due to premature study termination, the resulting sample size was not adequately powered to show superiority.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.